CLINICAL TRIAL: NCT06097143
Title: Performance of Flowable Giomer Versus Nanofilled Flowable Composite With or Without Giomer Coat In Conservative Occlusal Cavities: 18 Months Randomized Clinical Trial
Brief Title: Clinical Performance of Flowable Giomer Versus Nanofilled Composite in Conservative Occlusal Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amina Ahmed Abdellatif Hassan Gaafar, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Giomer Based Class I Cavities
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2023-11

CONDITIONS: Occlusal Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Flowable Giomer (Experimental): Patients with conservative carious class I occlusal cavities will be treated with Shofu™ Beautifil Injectable X, Shofu Dental Corp., Japan flowable composite Novel bio-active flowable resin containing nano S-PRG (Surface Pre-Reacted Glass ionomer).
  Interventions: Other: Flowable Giomer
- Nano-filled Flowable Composite with S-PRG barrier coat (Experimental): Patients with conservative carious class I occlusal cavities will be treated with Filtek™ Z350 XT 3M ESPE, USA Flowable composite: Conventional resin-based nano-filled flowable composite which will then be coated with Shofu™ PRG Barrier Coat, Shofu Dental Corp., Japan.
  Interventions: Other: Flowable Nano-filled composite with S-PRG barrier coat
- Nano-Filled Flowable Composite (Active Comparator): Patients with conservative carious class I occlusal cavities will be treated with Filtek™ Z350 XT 3M ESPE, USA Flowable composite: Conventional resin-based nano-filled flowable composite.
  Interventions: Other: Flowable Nano-filled composite

INTERVENTIONS:
Other: Flowable Giomer — Pre-reacted Glass Ionomer (PRG) filler is added to resin to create giomer, a dental adhesive material. Fluoride release and recharge, acid resistance, an anti-plaque effect, dentin remineralization, and acid buffering capacity are some of the benefits of giomer.
  Arms: Flowable Giomer
Other: Flowable Nano-filled composite with S-PRG barrier coat — Flowable composites are claimed to have a higher wetting ability of the tooth surface and thus ensure penetration into all surface irregularities in layers of minimal thickness. As a result of the higher amount of filler particles, it is noted that flowable composites have less porosity than conventional resin-based sealants. Moreover, flowable composite materials have better mechanical properties which lead to increased durability and longevity of the restoration.
  The PRG Barrier Coat is a resinous coating substance that shields the enamel surface from demineralization brought on by acidic attack. Near the coated surface, S PRG filler ions in PRG Barrier Coat have been found to have an acid-neutralizing effect. F and Sr released by PRG Barrier Coat can be effectively absorbed by the tooth substrate to prevent demineralization thus hindering the progression of caries.
  Arms: Nano-filled Flowable Composite with S-PRG barrier coat
Other: Flowable Nano-filled composite — Flowable composites are claimed to have a higher wetting ability of the tooth surface and thus ensure penetration into all surface irregularities in layers of minimal thickness. As a result of the higher amount of filler particles, it is noted that flowable composites have less porosity than conventional resin-based sealants. Moreover, flowable composite materials have better mechanical properties which lead to increased durability and longevity of the restoration.
  Arms: Nano-Filled Flowable Composite

SUMMARY:
With limited evidence-based information in literature the goal of this clinical trial is to learn about Flowable Giomer and compare it to Nanofilled Flowable Composite in Conservative Occlusal Cavities. It is beneficial to evaluate the newly introduced material using a randomized controlled clinical trial to test the null hypothesis that this new flowable giomer (Shofu™ Beautifil Injectable X, Shofu Dental Corp., Japan) and conventional resin-based nano-filled composite (Filtek™ Z350 XT 3M ESPE, USA) which will then be coated with (Shofu™ PRG Barrier Coat, Shofu Dental Corp., Japan) will have the same clinical performance as flowable resin composite as a preventative restorative restoration in permanent molars.

DETAILED DESCRIPTION:
This study will be conducted to clinically evaluate caries prevention and marginal integrity of flowable giomer and flowable resin composite coated with S-PRG in comparison to flowable resin composite as a preventative resin restoration in patients requiring minimally invasive simple class I cavities in permanent molars over 18 months test period.

Teeth that meet the inclusion criteria will be selected. The occlusal surfaces will be cleaned by pumice and a low speed polishing brush. Baseline recording of carious lesions will be carried out using DIAGNOdent pen. Cavity preparation will be carried out using number 330 (Mani, Inc., Japan) bur.

All the tested materials Shofu™ Beautifil Injectable X, (Shofu Dental Corp., Japan flowable composite) and Filtek™ Z350 XT (3M ESPE, USA) Flowable composite: Conventional resin-based nano-filled flowable composite which will then be coated with Shofu™ PRG Barrier Coat, (Shofu Dental Corp., Japan) will be used according to manufacturer instructions and comparator restorative material Filtek™ Z350 XT (3M ESPE, USA) Flowable composite.

All restorations will be finished using flame-shaped finishing stone (Mani, Inc., Japan) and polished using rubber cups (Kerr Corporation, Orange, CA, USA).

The primary and secondary outcomes will be measured at four intervals 1 week after placement, 6 months follow up, 12 months follow up and 18 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or Bilateral small Class I carious lesions
* Patients with good oral health
* Small Class I carious lesion in occlusal pits and fissures

Exclusion Criteria:

* Existing systemic diseases
* Severe medical complications
* Allergy history concerning methacrylates
* Pregnancy
* Heavy smoking
* Evidence of severe bruxism, clenching or temporomandibular joint disorders
* Presence of existing occlusal restoration
* Periapical or pulpal pathology
* Tooth hypersensitivity
* Possible prosthodontic restoration of teeth
* Endodontically treated teeth
* Severe periodontal affection

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-21 (Actual)

PRIMARY OUTCOMES:
Fracture and Retention of Material | T0= 1 week postoperative T1= 6 months follow up T2= 12 months follow up T3= 18 months follow up
  World Dental Federation (FDI) criteria (Hickel et al.,2010) Scores:
  1. Clinically excellent/ very good 1.1 No fractures/cracks
  2. Clinically good 2.1 Small hairline crack
  3. Clinically sufficient/ satisfactory 3.1 Two or more larger hairline cracks and/or material chip not affecting the marginal integrity or approximal contact
  4. Clinically unsatisfactory (but repairable) 4.1 Material chip fractures which damage marginal quality or approximal contacts 4.2 Bulk fractures with partial loss (less than half of the restoration)
  5. Clinically poor (replacement necessary) 5.1 Partial or complete loss of restoration or multiple fractures

SECONDARY OUTCOMES:
Occlusion and wear | T0= 1 week postoperative T1= 6 months follow up T2= 12 months follow up T3= 18 months follow up
  World Dental Federation (FDI) criteria
Marginal Adaptation | T0= 1 week postoperative T1= 6 months follow up T2= 12 months follow up T3= 18 months follow up
  World Dental Federation (FDI) criteria
Form and contour | T0= 1 week postoperative T1= 6 months follow up T2= 12 months follow up T3= 18 months follow up
  World Dental Federation (FDI) criteria
Dental hard tissue defects at restoration margins | T0= 1 week postoperative T1= 6 months follow up T2= 12 months follow up T3= 18 months follow up
  World Dental Federation (FDI) criteria
Postoperative hypersensitivity/pulp status | T0= 1 week postoperative T1= 6 months follow up T2= 12 months follow up T3= 18 months follow up
  World Dental Federation (FDI) criteria
Incidence of new carious lesions | T0= 1 week postoperative T1= 6 months follow up T2= 12 months follow up T3= 18 months follow up
  Intra-oral quantitative light-induced fluorescence applied on the occlusal surface of permanent molars with initial Class I caries using DIAGNOdent pen
  Scores:
  0 - 14 indicate a healthy occlusal surface 15 - 20 indicate the presence of enamel caries, 21 or more indicate the presence of dentinal caries

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogawa Y, Sayed M, Hiraishi N, Al-Haj Husain N, Tagami J, Ozcan M, Shimada Y. Effect of Surface Pre-Reacted Glass Ionomer Containing Dental Sealant on the Inhibition of Enamel Demineralization. J Funct Biomater. 2022 Oct 14;13(4):189. doi: 10.3390/jfb13040189. PMID 36278658
- [Background] Baroudi K, Rodrigues JC. Flowable Resin Composites: A Systematic Review and Clinical Considerations. J Clin Diagn Res. 2015 Jun;9(6):ZE18-24. doi: 10.7860/JCDR/2015/12294.6129. Epub 2015 Jun 1. PMID 26266238
- [Background] Jafarzadeh M, Malekafzali B, Tadayon N, Fallahi S. Retention of a Flowable Composite Resin in Comparison to a Conventional Resin-Based Sealant: One-year Follow-up. J Dent (Tehran). 2010 Winter;7(1):1-5. Epub 2010 Mar 31. PMID 21998768
- [Background] Asefi S, Eskandarion S, Hamidiaval S. Fissure sealant materials: Wear resistance of flowable composite resins. J Dent Res Dent Clin Dent Prospects. 2016;10(3):194-9. doi: 10.15171/joddd.2016.031. Epub 2016 Aug 17. PMID 27651887
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Jaafar N, Ragab H, Abedrahman A, Osman E. An In Vivo Investigation of Diagnostic Performance of DIAGNOdent Pen and the Canary System for Assessment and Monitoring Enamel Caries under Fissure Sealants. J Int Soc Prev Community Dent. 2020 Jun 15;10(3):246-254. doi: 10.4103/jispcd.JISPCD_480_19. eCollection 2020 May-Jun. PMID 32802769
- [Background] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2573-2592. doi: 10.1007/s00784-022-04814-1. Epub 2022 Dec 12. PMID 36504246
- [Background] Kawasaki K, Kambara M. Effects of ion-releasing tooth-coating material on demineralization of bovine tooth enamel. Int J Dent. 2014;2014:463149. doi: 10.1155/2014/463149. Epub 2014 Jan 21. PMID 24578706
- [Background] Funato Y, Matsuda Y, Okuyama K, Yamamoto H, Komatsu H, Sano H. A new technique for analyzing trace element uptake by human enamel. Dent Mater J. 2015;34(2):240-5. doi: 10.4012/dmj.2014-127. Epub 2015 Feb 25. PMID 25740308
- [Background] Shaalan OO, Abou-Auf E, El Zoghby AF. Clinical evaluation of flowable resin composite versus conventional resin composite in carious and noncarious lesions: Systematic review and meta-analysis. J Conserv Dent. 2017 Nov-Dec;20(6):380-385. doi: 10.4103/JCD.JCD_226_17. PMID 29430087